CLINICAL TRIAL: NCT04829110
Title: Alcohol Induced de Novo Lipogenesis in Women
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Justin Fletcher, Assistant Professor, University of Texas Southwestern Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: STU-2021-0246
Record Dates: First submitted 2021-03-18; First posted 2021-04-02 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-03

CONDITIONS: Liver Metabolism
MeSH Terms: interventions — Sucrose; sodium lactobionate sucrose solution

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- A. ETOH (Experimental): 5 Males and 5 Females will receive deuterated water and drink 2.15 ounces of alcohol in the form of vodka and have de novo Lipogenesis measured at 11 time points during and after.
  Interventions: Other: ETOH
- ETOH + Sucrose (Experimental): 5 Females will receive deuterated water and drink 1.72 ounces of alcohol in the form of vodka + 7 grams of sucrose and have de novo Lipogenesis measured at 11 time points during and after.
  Interventions: Other: ETOH; Other: Sucrose
- C. Sucrose (Experimental): 5 Females will receive deuterated water and drink a solution containing water and 35 grams of sucrose, and have de novo Lipogenesis measured at 11 time points during and after.
  Interventions: Other: Sucrose

INTERVENTIONS:
Other: ETOH — Participants will consume Vodka
  Other Names: Vodka
  Arms: A. ETOH; ETOH + Sucrose
Other: Sucrose — Participants will consume sucrose in solution with water
  Other Names: Sucrose solution
  Arms: C. Sucrose; ETOH + Sucrose

SUMMARY:
The study is cross-sectional is design. In the first Aim of this study, 5 women and 5 men will be asked to consume 2g/kg of [2H]water (a.k.a. deuterium oxide or heavy water) which incorporates 2H tracers into newly synthesized fatty acids and triglycerides. Deuterated water is not radioactive and has a long history of application in human studies. Researchers will collect blood samples 2 hours before and 5 hours after the participants consume 20 grams of alcohol as vodka to measure alcohol induced hepatic de novo lipogenesis (DNL) in both men in women. In addition, for Aim 2 researchers will recruit an additional 10 women who will be randomized into one of two groups who will consume a beverage containing vodka and sucrose, or sucrose alone. Aim 2 will be identical to the experimental scheme in Aim 2 in order to determine if sucrose enhances the effects of vodka on hepatic DNL.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female
* Ages 21 - 45
* Healthy
* Light to moderate alcohol consumption (≤1 drink a day (~14g) in women and ≤2 drinks a day (~28 g) in men)
* BMI between 18.5-29.9
* Normal Nutritional Status
* Ability to speak and understand English

Exclusion Criteria:

* BMI >29.9
* Comorbid conditions
* Any regular medications, except Oral Contraceptives
* Pregnant or Breastfeeding
* Regular exercise above activities of daily living

Ages: 21 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2021-11-11 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Mean Change in Hepatic De Novo Lipogenesis (DNL) | 0, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, and 7 hours post heavy water consumption
  DNL will be measured by Orbitrap high-resolution-mass-spectrometry (GC-Orbitrap-HRMS)
  We will measure changes in the incorporation of 2H tracers into plasma triglycerides over time. This data will be analyzed by averaging each time point and looking at change in de novo lipogenesis over time.

CONTACTS AND LOCATIONS:
Locations (1):
- School of Health Professions at UTSW, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No